CLINICAL TRIAL: NCT02577536
Title: PregSource: Crowdsourcing to Understand Pregnancy, Observations of Daily Living From Pregnant Women
Brief Title: PregSource: Crowdsourcing to Understand Pregnancy
Acronym: PregSource
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PregSource; NCT02659969 (obsolete NCT alias)
Record Dates: First submitted 2015-10-05; First posted 2015-10-16 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy; Pregnancy Complications; Morning Sickness; Diabetes, Gestational; Placenta Diseases; Birth Weight
Keywords: Pregnancy outcome; Neonatal outcome; Birth weight; Weight gain; Physical disability
MeSH Terms: conditions — Pregnancy Complications; Morning Sickness; Diabetes, Gestational; Placenta Diseases; Birth Weight; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 All Subjects: No interventions
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No Interventions will be conducted under this study.

SUMMARY:
PregSource uses a crowd-sourcing approach, asking pregnant women to enter information regularly and directly about their pregnancies throughout gestation and the early infancy of their babies into online surveys and trackers via a website and/or mobile application ("app"). In exchange, participants can track their data over time, print out reports to share with their healthcare team, and see how they compare to other women. In addition, PregSource will provide participants with links to trusted, evidence-based information about pregnancy management, issues, and complications.

More information is available at: https://pregsource.nih.gov

DETAILED DESCRIPTION:
The objective of PregSource: Crowdsourcing to Understand Pregnancy (PregSource) is: to better understand the range of physical and emotional experiences and alterations in behavior that women have during pregnancy and after giving birth, the impact of these experiences on women's lives, and the perinatal challenges encountered by special sub-populations of women.

PregSource uses a longitudinal, crowd-sourcing, citizen science approach, asking pregnant women regularly and directly about their pregnancies. Participants enter information throughout gestation and the early infancy of their babies into online surveys and trackers via a website and/or mobile application ("app"). In exchange, participants will be able to track their pregnancy data over time, print out reports to share with their healthcare team, and view summaries of de-identified data to see how they compare to other women. In addition, PregSource will provide participants with links to trusted, evidence-based information from partner organizations about pregnancy management, issues, and complications.

Participants may also be a potential pool of recruits for clinical studies. Based on information they enter, eligible women who are interested in participating in clinical studies may be sent contact information about observational or interventional studies. Their contact information will not be shared directly with researchers.

After a critical mass of data is collected, de-identified data will be available to approved researchers for analysis.

If you are pregnant and interested in joining PregSource, please:

1. Go to https://pregsource.nih.gov/.
2. Select "Join" at the top of the page.
3. Complete the questions on the Join page
4. Complete the online consent form.

After that you will be asked some information for your account Profile, and you should start receiving/seeing questionnaires to complete on the My Dashboard page. You can also come in as often as you want/need to to complete PregSource's trackers to tell us about your mood, activity level, sleep, morning sickness, and weight gain. We also have a separate tracker for adding any medications, vitamins, and other supplements you may take during your pregnancy.

More information is available at: https://pregsource.nih.gov. If you have any additional questions, please let us know at pregsource@nih.gov.

ELIGIBILITY:
Inclusion Criteria:

* Women who are pregnant

Exclusion Criteria:

* Males
* Women who are not pregnant
* Women under 18 years of age or older than 70 years of age
* Women who are unable to provide consent for themselves, and for whom a parent, legal guardian, or legally authorized representative does not provide consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All pregnancy women 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 2359 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of women delivering at each gestational week | Up to 44 weeks gestational age
  Gestational age at pregnancy end date

SECONDARY OUTCOMES:
Birthweight of baby | At delivery
  Birthweight of babies born >20 weeks gestational age
Maternal weight gain in pregnancy by gestational age | Up to 44 weeks gestational age
  Maternal weight gain in pregnancy by gestational age
Number of women without pregnancy complications | Up to 44 weeks gestational age
  Pregnancy complications including: gestational diabetes, preeclampsia, placenta previa, etc.)
Number of live births | At birth
  Number of infants born alive

CONTACTS AND LOCATIONS:
Overall Officials: Caroline C Signore, MD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Melissa Parisi, MD PhD, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited into the NICHD data repository.
Supporting Information: Study Protocol, ICF
Time Frame: Deposited by August 31, 2023
Access Criteria: Per NICHD's Data and Specimen Hub (DASH) policy
URL: https://dash.nichd.nih.gov/

REFERENCES:
- See also: PregSource home page — https://pregsource.nih.gov
- Available data/document: Individual Participant Data Set — https://dash.nichd.nih.gov/study/424642 — Deidentified data from this study are not available in the NICHD Data and Specimen Repository.

DOCUMENTS (2):
  • Study Protocol (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT02577536/Prot_000.pdf
  • Informed Consent Form (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT02577536/ICF_001.pdf